CLINICAL TRIAL: NCT02316782
Title: Bifurcation Lesion Analysis and STenting / BLAST
Acronym: BLAST
Status: Completed | Type: Observational
Sponsor: Volcano Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: RSC-001
Record Dates: First submitted 2014-05-14; First posted 2014-12-15 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Coronary Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-blinded IVUS assessment: The non-blinded arm will use the angiogram and IVUS grayscale and VH-IVUS to guide the procedure.
  Interventions: Device: Nonblinded IVUS
- Blinded IVUS assessment: After routine coronary angiogram, the physicians in the blinded arm of the study will only use the angiogram to guide the DES stenting procedure;
  Interventions: Device: Blinded IVUS assessment

INTERVENTIONS:
Device: Blinded IVUS assessment — Only the angiogram is used for stent placement
  Groups: Blinded IVUS assessment
Device: Nonblinded IVUS — Angiogram, Grayscale IVUS and VH IVUS used for stent placement pre and post intervention
  Groups: Non-blinded IVUS assessment

SUMMARY:
The purpose of this research study is to determine if Intravascular Ultrasound (IVUS) grayscale and VH (Virtual Histology)-IVUS pre-stenting can assess more accurately the location, amount, and type of a blockage than angiogram alone. Additionally, this study is to determine if IVUS grayscale and VH-IVUS guidance will result in improved acute and long term procedural outcome vs. bifurcation stenting with only angiographic guidance in native coronary arteries.

DETAILED DESCRIPTION:
Global multi-center, prospective, two-arm, randomized study. Patients will be randomized to either blinded or non-blinded IVUS assessment before the treatment of coronary bifurcation lesions. Treatment will be based either on grayscale and VH IVUS versus angiography alone.

After routine coronary angiogram, the physicians in the blinded arm of the study will only use the angiogram to guide the DES stenting procedure; the non-blinded arm will use the angiogram and IVUS grayscale and VH-IVUS to guide the procedure. In all patients, both pre- and post intervention, IVUS grayscale and VH-IVUS will be preformed on both branches of the bifurcation (blinded or non-blinded).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be greater than 18 years of age.
2. Patient is scheduled for coronary stenting of a bifurcation lesion in a native artery using Drug Eluting Stents (DES).
3. Patient must be willing and able to read and sign the informed consent document before planned coronary intervention.
4. If the patient is female and of child bearing potential, a pregnancy test (serum HcG or urine dip stick) is negative within 7 days of the procedure.
5. Side branch lumen diameter min of >2 mm by visual, angiographic estimate.
6. Patient must agree to be available for follow-up at 30 days, 1 and 2 years after procedure.
7. Other significant lesions in different vessels should be treated successfully (residual stenosis < 30%, normal TIMI flow, no EKG modification) before treating the index bifurcation lesion.

   -

Exclusion Criteria:

1. The patient experiences significant hepatic disease, renal disease, lung disease and/or malignant disease with unfavorable prognosis.
2. Any contraindications for IVUS interrogation as determined by the investigator including sever vessel tortuosity and severe calcification by angiogram.
3. Side branch lumen diameter < 2 mm by visual, angiographic estimate.
4. The patient suffered a cerebrovascular accident within the past 6 months and has residual effects from the event.
5. The patient suffered significant (as determined by the Investigator) gastrointestinal bleeding within the past 3 months.
6. The most recent white blood cell count less than 3,000 cell/mm3 or the number of platelet is less than 100,000 cell/mm3.
7. The patient has contraindication to antithrombotic regimen or anticoagulation therapy.
8. Any other patients who are judged by principal Investigator to be inappropriate for participation in the trial.
9. Existing hemorrhagic disease or coagulation problems creating inability to obtain homeostasis at entry site.
10. The patient has history of or known reaction or sensitivity to contrast agent and is unable to be premedicated.
11. Hemodynamic instability at the time of intervention.
12. Severe chronic renal insufficiency (plasma/ serum creatinine > 2.5mg/dl) at the time of intervention, except for patients on dialysis.
13. The lesion is 0.0.1. (Medina classification).
14. The bifurcation lesion involves an anastamosis site from previous a coronary artery bypass surgery.
15. Acute MI or recent MI with CPK > 3 times the normal value prior to intervention (during index hospitalization).
16. Other significant lesion in the same vessel.
17. Other lesion in a different vessel not successfully treated

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Per Protocol Population All patients who met all inclusion/exclusion criteria, completed the study intervention procedure as described in the protocol, and completed the 1-month follow-up.
  Intent to Treat Any subject randomized into the trial and there was an attempt to use the IVUS but either side branch was not IVUS'd pre and post intervention.
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2008-10; Primary Completion 2010-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
IVUS with VH guidance leads to better post procedural outcomes when compared | 2 years
  The primary objective of this randomized study is to demonstrate that pre-intervention IVUS can provide more accurate information on lesion characteristics than information derived from pre-procedural angiogram alone. This will be determined by full lesion coverage, no acute evidence of plaque protrusion or dissection at the stent edge, no evidence of stent underexpansion, no evidence of stent malapposition, or no significant side branch disease left behind.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lefevre, M.D., Principal Investigator — Institute Hospitalier J Cartier
Locations (10):
- Saint Luke's Hospital-Mid America Heart Institute, Kansas City, Missouri, United States
- Kardiologisk laboratorium/B-lab Skejby Sygehus, Aarhus, Denmark
- France (3):
  - Clinique Saint Augustin, Bordeaux
  - Hopital de la Cavale Blanche-CHU, Brest
  - Nouvelles Cliniques Nantaises, Nantes
- Azienda Sanitaria Ospedaliera Molinette San Giovanni Battista al Torino Departp Emodinamica Universitaria, Torino, Italy
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Medisch Spectrum Twente, Enschede, Netherlands
- CSK MSWiA w Warszawie, Warsaw, Poland
- St. Thomas Hospital Cardiothoracic Centre, London, United Kingdom